CLINICAL TRIAL: NCT06758297
Title: Effect of Artificial Intelligence-Assisted Motivational Talk on Patients' Fear of Movement and Mobility Level After Knee Replacement: a Randomized Controlled Trial
Brief Title: Effect of Artificial Intelligence-Assisted Motivational Talk on Patients' Fear of Movement and Mobility Level After Knee Replacement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Hatice Merve Alptekin, research assistant, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025/01
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Knee Arthroplasty, Total

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-Powered Motivational Speech Group (Experimental): 1. Patients will be assessed for fear of falling using the "Descriptive Characteristics Form" and the "TAMPA Kinesiophobia Scale".
  2. The audio recording prepared with artificial intelligence support will be listened to 3 times.
  4. . Patients will be assessed for fear of falling again using the "TAMPA Kinesiophobia Scale".
  5. While the patients are standing up, the researcher will measure their mobility levels using the "Patient Mobility and Observer Mobility Scale".
  Interventions: Other: AI-Powered Motivational Speech
- Control Group (No Intervention): 1. Patients will be assessed for fear of falling using the "Descriptive Characteristics Form" and the "TAMPA Kinesiophobia Scale".
  2. After 15 minutes, patients will be assessed for fear again using the "TAMPA Kinesiophobia Scale".
  3. While the patients are being stood up, the researcher will measure their mobility levels using the "Patient Mobility and Observer Mobility Scale".

INTERVENTIONS:
Other: AI-Powered Motivational Speech — It is known that patients with knee prosthesis have difficulty in the first standing process due to fears of falling, not being able to walk again, and recurrence of their disease. For this purpose, a speech text that will motivate patients was prepared with the support of "ChatGPT". Expert opinions were obtained from 2 orthopedic specialists and 2 specialist psychiatric nurses for this speech text. Later, the speech text was converted into an audio video with the "ElevenLabs" application. Thus, it was planned to make it easier for patients to listen to it again. Patients will listen to this motivational speech in their own patient rooms and using their own headphones.
  Arms: AI-Powered Motivational Speech Group

SUMMARY:
Patients may have fears about moving after TKA surgery. This fear has been described in the literature. Fear of re-injury has also been called kinesiophobia, which is the primary psychosocial structure in the fear-avoidance model. Injury or surgery can create feelings of uncertainty and fear of how much the injury will affect future function. This situation causes the individual to have negative attitudes towards activity. For this reason, kinesiophobia is a psychological element that can affect patient outcomes and recovery after knee trauma or knee surgery. Kinesiophobia is considered a normal reaction in the early postoperative period. However, it can affect patients' early mobility after TKA. It is important to improve functional outcomes in the early period, especially in knee surgeries. Patients may delay mobilization because they feel a fear of falling after surgery, and as this delay increases, their mobility is affected worse. The only solution to this situation, which can enter a vicious circle, is to determine patients' fear of falling and apply interventions accordingly. There are studies in the literature evaluating the fear of movement after total knee arthroplasty and its effect on patients' mobility levels. However, no study has been found investigating the effect of a motivational speech prepared with the help of artificial intelligence on patients. The World Health Organization (WHO) has published a four-year global strategy report on digital health within the scope of the vision of health everywhere and for everyone. According to this report, digital health is defined as "the adoption of digital technologies to improve and develop health". The use of artificial intelligence technology is increasing day by day in the changing and developing world. It is known that nurses constitute 45% of all health professionals in the field of health and that insufficient staff number continues to be a priority problem. It is expected that insufficient staff will be supported and efficiency will increase with the contribution of artificial intelligence, which is the copy of human intelligence with advanced technology. With this research, we aim to both support staff and improve patient outcomes by using artificial intelligence technologies. The aim of this study is to evaluate the effect of an artificial intelligence-supported motivational speech on patients' fear of movement and mobility level after knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have had knee replacement surgery,
* Be over 18 years of age,
* Agree to participate in the study,
* Be able to understand and speak Turkish,
* Be able to read and write

Exclusion Criteria:

* Cancellation or postponement of patient's surgery
* Patients in pain,
* Those whose walking is not recommended by the physician,
* Those with mental disabilities or psychological disorders,
* Patients who are alcohol or drug addicts,
* Those with hearing or visual impairments,
* Patients who do not want to use the headphones that will be used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Kinesiophobia | 20 minutes before the patient starts walking, 5 minutes before the patient starts walking
  The patients' fear of falling will be evaluated with the TAMPA Kinesiophobia Scale. The scale is a 17-question scale developed to determine the level of injury/re-injury and fear-avoidance processes related to activities. The scale is scored with a four-point Likert scoring type of "1=Strongly Disagree", "2=Disagree", "3=Agree", "4=Strongly Agree". The minimum score value obtained from the scale is 17, while the maximum score value is 68. Vlaeyen et al. accepted a score above 37 from the scale as a high level of kinesiophobia.

SECONDARY OUTCOMES:
Mobility Level | Simultaneously when the patient first stands up (approximately the 2nd postoperative day)
  The patient's mobility will be assessed with the Patient Mobility and Observer Mobility Scales. The scale is a 5-point Likert-type scale with a 5-point score ranging from "It was very easy" to "It was very difficult". In the Mobility Scale, the dependency/independence status/degree during the performance of four activities after surgery is numbered between 1 and 5. A score of 1 indicates that the patient performed the relevant activity independently without verbal warning or physical assistance, and a score of 5 indicates that the patient could not perform the relevant activity despite verbal warning or physical assistance. The total score is calculated by adding the scores for turning, sitting, standing and walking. A total score of 4-20 is obtained from the scale. An increase in the score indicates that the patient's movement skills are inadequate, and a decrease in the score indicates that their movement skills after the surgical intervention are good/sufficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun Gazi State Hospital, Samsun, Samsun, Turkey (Türkiye)